CLINICAL TRIAL: NCT07061717
Title: A Phase III, Randomized, Open-Label Clinical Trial Comparing Endocrine Therapy Combined With High-Dose Palbociclib and Hydroxychloroquine to Endocrine Therapy Combined With Standard-Dose Palbociclib for Hormone Receptor-Positive and HER2-Negative Advanced Breast Cancer
Brief Title: Comparing Endocrine Therapy Combined With High-Dose Palbociclib and Hydroxychloroquine to Endocrine Therapy Combined With Standard-Dose Palbociclib for Hormone Receptor-Positive and HER2-Negative Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chang Gong, professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2025-424-01
Record Dates: First submitted 2025-05-28; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Hormone Receptor-Positive and HER2-Negative Advanced Breast Cancer
MeSH Terms: interventions — palbociclib; Anastrozole; Letrozole; exemestane; Hydroxychloroquine; BID protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group1 (Active Comparator): Standard-Dose Palbociclib + Endocrine therapy
  Interventions: Drug: Palbociclib 125mg qd (3 weeks of treatment followed by 1 week off) + Anastrozole 1mg qd / Letrozole 2.5mg qd / Exemestane 25mg qd
- Experimental Group 1 (Experimental): Standard-Dose Palbociclib + Endocrine Therapy + Hydroxychloroquine
  Interventions: Drug: Palbociclib 125mg qd (3 weeks of treatment followed by 1 week off) + Anastrozole 1mg qd / Letrozole 2.5mg qd / Exemestane 25mg qd + Hydroxychloroquine 600mg bid
- Experimental Group 2 (Experimental): High-Dose Palbociclib + Endocrine Therapy + Hydroxychloroquine
  Interventions: Drug: Palbociclib 200mg qd (3 weeks of treatment followed by 1 week off) + Anastrozole 1mg qd / Letrozole 2.5mg qd / Exemestane 25mg qd + Hydroxychloroquine 600mg bid

INTERVENTIONS:
Drug: Palbociclib 125mg qd (3 weeks of treatment followed by 1 week off) + Anastrozole 1mg qd / Letrozole 2.5mg qd / Exemestane 25mg qd — Standard-Dose Palbociclib + Endocrine therapy
  Arms: Control Group1
Drug: Palbociclib 125mg qd (3 weeks of treatment followed by 1 week off) + Anastrozole 1mg qd / Letrozole 2.5mg qd / Exemestane 25mg qd + Hydroxychloroquine 600mg bid — Standard-Dose Palbociclib + Endocrine Therapy + Hydroxychloroquine
  Arms: Experimental Group 1
Drug: Palbociclib 200mg qd (3 weeks of treatment followed by 1 week off) + Anastrozole 1mg qd / Letrozole 2.5mg qd / Exemestane 25mg qd + Hydroxychloroquine 600mg bid — High-Dose Palbociclib + Endocrine Therapy + Hydroxychloroquine
  Arms: Experimental Group 2

SUMMARY:
This is a a phase III, randomized, open-label clinical trial comparing endocrine therapy combined with high-dose palbociclib and hydroxychloroquine to endocrine therapy combined with standard-dose palbociclib for hormone receptor-positive and her2-negative advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria :

1. Voluntary participation in this study and signed informed consent.
2. Female (aged ≥18 and ≤70 years), histologically or cytologically diagnosed as HER2-negative (based on ASCO/CAP guidelines: HER2 IHC 2+/FISH negative, IHC 1+ or IHC 0), hormone receptor-positive (based on ASCO/CAP guidelines: ER ≥1%) breast cancer, with evidence of locally recurrent or metastatic disease that is not suitable for surgical resection or curative radiotherapy.
3. Locally recurrent or metastatic breast cancer that has not received any prior systemic anticancer treatment.
4. Presence of measurable lesions according to RECIST v.1.1, or isolated bone lesions. Tumor lesions previously treated with radiation or other local therapies are considered measurable only if disease progression at the treated site is clearly documented after completion of therapy.
5. ECOG performance status of 0-1.
6. Sufficient bone marrow function reserve: white blood cell count ≥3.0×10⁹/L, neutrophil count ≥1.5×10⁹/L, platelet count ≥100×10⁹/L, hemoglobin ≥90 g/L.
7. Sufficient liver and kidney function reserve: AST and ALT ≤3 times the upper limit of normal (5 times in the case of liver metastasis), total bilirubin ≤1.5 times the upper limit of normal (3 times in case of Gilbert's syndrome), serum creatinine and urea nitrogen ≤1.5 times the upper limit of normal.
8. All acute toxicities from prior anticancer treatments or surgical interventions have resolved to ≤Grade 1 according to NCI-CTCAE v.5.0 (alopecia or other toxicities that are not considered to pose a safety risk, in the investigator's judgment, are exceptions).
9. Willing and able to comply with scheduled visits.

Exclusion Criteria :

1. Presence of complications that the investigator considers may become life-threatening in the short term (including massive effusions (pleural effusion, pericardial effusion, ascites), carcinomatous lymphangitis, liver involvement exceeding 50%).
2. Known, uncontrolled clinical symptoms, brain edema and/or progressive growth of symptomatic central nervous system metastases, carcinomatous meningitis, or meningeal disease.
3. Any major surgery, chemotherapy, radiotherapy, any investigational drug or other anticancer treatments within 2 weeks prior to randomization. Patients who have received >25% bone marrow irradiation, regardless of the timing of the radiotherapy, are excluded.
4. Diagnosis of any other malignancy within 3 years prior to randomization, except for adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, or cervical carcinoma in situ.
5. QTc >480 milliseconds (based on electrocardiogram), or a family or personal history of long QT syndrome, short QT syndrome, Brugada syndrome, or known QTc prolongation, or history of Torsades de Pointes (TdP).
6. Presence of uncontrolled electrolyte disturbances that may exacerbate the effects of QTc prolonging drugs (e.g., hypocalcemia, hypokalemia, hypomagnesemia).
7. Within 6 months after randomization, the occurrence of any of the following: myocardial infarction, severe/uncontrolled angina, NCI-CTCAE v.5.0 Grade 2 persistent arrhythmias, any degree of atrial fibrillation, coronary/peripheral artery bypass surgery, asymptomatic congestive heart failure, cerebrovascular accident (including transient ischemic attack), or asymptomatic pulmonary embolism.
8. Active inflammatory bowel disease, chronic diarrhea, short bowel syndrome, or any upper gastrointestinal surgery (including gastrectomy).
9. Known allergy to anastrozole, letrozole, exemestane/hydroxychloroquine/palbociclib, or any excipients of these agents.
10. Known human immunodeficiency virus infection.
11. Participation in another clinical study involving investigational drugs during the active treatment phase of this trial.
12. Positive for HBV surface antigen with high HBV DNA copy number (except for those with low copy number (≤103/ml) after antiviral treatment).
13. Ophthalmologic examination revealing any of the following eye conditions: retinopathy, visual field defects, etc.
14. Any other severe acute or chronic medical or psychiatric conditions, or laboratory abnormalities, which may increase the risk associated with participation in the study or the use of the investigational product, or which may interfere with the interpretation of study results, and in the investigator's judgment, would make the patient unsuitable for participation in the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) as Assessed by the Investigator | 3 years after random assignment

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) as Assessed by Blinded Independent Central Review (BICR) | 3 years after random assignment
Overall Survival (OS) | 3 years after random assignment
Objective Response Rate (ORR) | 3 years after random assignment
Clinical Benefit Rate (CBR) | 6 months after random assignment
Treatment Associated Adverse Effect | 3 years after random assignment
Patient-Reported Outcomes (PRO) | 3 years after random assignment

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No